CLINICAL TRIAL: NCT06432933
Title: Comparison of Apnea-Hypopnea Index, in Patients With Potentially Undiagnosed Obstructive Sleep Apnea, Treated With or Without Preventive Oxygen Therapy, During the First Night After Bariatric Surgery
Brief Title: Comparison of Apnea-Hypopnea Index in Patients With or Without Preventive Oxygen Therapy After Bariatric Surgery
Acronym: OXYBAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-2352
Record Dates: First submitted 2024-04-03; First posted 2024-05-29 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Obstructive Sleep Apnea; Obesity; Bariatric Surgery Candidate
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Without preventive oxygen therapy (Experimental)
  Interventions: Other: No preventive oxygen therapy (2L)
- With preventive oxygentherapy (Active Comparator)
  Interventions: Other: Preventive oxygen therapy (2L) standard care

INTERVENTIONS:
Other: No preventive oxygen therapy (2L) — Participants will not receive preventive oxygen 2L during the first postoperative night after bariatric surgery.
  Arms: Without preventive oxygen therapy
Other: Preventive oxygen therapy (2L) standard care — Participants will receive preventive oxygen 2L during the first postoperative night after bariatric surgery, standard care.
  Arms: With preventive oxygentherapy

SUMMARY:
The best perioperative strategy for obstructive sleep apnea (OSA) in bariatric surgery remains unclear. A strategy is to monitor patients and administer preventive oxygen therapy during the first postoperative night. However it is unknown what if preventive oxygen therapy is necessary.

The goal of this trial is to compare the Apnea-Hypopnea Index (AHI) in participants with or without preventive oxygen therapy.

Methods:

Participants are patients who underwent bariatric surgery without treated OSA and will be will be randomized into arm A or arm B:

Arm A: First postoperative night in the hospital with preventive oxygen therapy (standard care), Arm B: First postoperative night in hospital without preventive oxygen therapy (intervention).

DETAILED DESCRIPTION:
Rationale: The prevalence of obstructive sleep apnea (OSA) in the bariatric surgery population is high and mostly undiagnosed. The best perioperative strategy to manage sleep apnea in bariatric patients remains unclear. A recent study found that monitoring patients with pulsoximetry and giving them preventive oxygen therapy during the first postoperative night is safe and cost effective. In a population with patients with OSA but without obesity, no significant difference in apnea hypopnea index (AHI) was found between patients with and without oxygen therapy during the first postoperative night. The question was raised if preventive oxygen therapy during the first postoperative night after bariatric surgery is needed.

Objective: The primary objective of this study is to compare AHI in patients with potentially undiagnosed OSA, treated with or without preventive oxygen therapy, during the first night after bariatric surgery. The secondary objective of this study is to compare sleep architecture in these patients

Study design: This is a randomized controlled non-inferiority trial consisting of two arms; Arm A: First postoperative night in the hospital with preventive oxygen therapy (standard care), Arm B: First postoperative night in hospital without preventive oxygen therapy (intervention).

Study population: Patients scheduled for primary bariatric surgery without treated OSA Intervention: During the first postoperative night at the hospital patients in intervention arm B will not receive preventive oxygen therapy.

Main study parameters/endpoints: Primary endpoint is AHI and secondary endpoints are 30 days complications rate, nursing intervention rate and parameters for sleep architecture and sleep related breathing, score of the Epworth Sleepiness Scale (ESS) and STOP BANG.

ELIGIBILITY:
Inclusion Criteria:

* Undergo primary bariatric surgery (RYGB or SG)
* Speak and read the Dutch language

Exclusion Criteria:

* Revisional bariatric surgery (e.g. sleeve conversion, RYGB after gastric banding)
* Same-day discharge after bariatric surgery
* Diagnosed OSA with treatment (CPAP, oral appliances)
* Professional drivers
* Use of alpha blockers
* Unable to speak or read the Dutch language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2024-04-09 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
Apnea-Hypopnea Index (AHI) | First postoperative night
  AHI will be measured by a home sleep study device (Watchpat300) and will be compared between both arms, the higher the AHI the more severe the sleep apnea

SECONDARY OUTCOMES:
Complication rate | Until 30 days after surgery
  All complication will be scored and will be compared between both arms
The number of nursing interventions | First postoperative night
  Nursing interventions will be scored on a form and the number of nursing interventions will be compared between both arms
Type of nursing interventions | First postoperative night
  e.g. waking up the patient or starting or increasing oxygen therapy/flow, this will be compared between both arms.
Oxygen Desaturation Index (ODI) | First postoperative night
  ODI will be measured by a home sleep study device (Watchpat300) and will be compared between both arms
AHI during Rapid Eye Movement (REM) sleep | First postoperative night
  AHI during REM sleep will be measured by a home sleep study device (Watchpat300) and will be compared between both arms
Respiratory disturbance index (RDI) | First postoperative night
  RDI will be measured by a home sleep study device (Watchpat300) and will be compared between both arms
Mean saturation | First postoperative night
  Mean saturation will be measured by a home sleep study device (Watchpat300) and will be compared between both arms
Mean saturation during desaturations, | First postoperative night
  Mean saturation during desaturations will be measured by a home sleep study device (Watchpat300) and will be compared between both arms
Number of desaturations | First postoperative night
  Number of desaturations will be measured by a home sleep study device (Watchpat300) and will be compared between both arms
Percentage of saturation <90% | First postoperative night
  will be measured by a home sleep study device (Watchpat300) and will be compared between both arms
Percentage of saturation <88% | First postoperative night
  will be measured by a home sleep study device (Watchpat300) and will be compared between both arms
Percentage of saturation <85% | First postoperative night
  will be measured by a home sleep study device (Watchpat300) and will be compared between both arms
Percentage of saturation <80% | First postoperative night
  will be measured by a home sleep study device (Watchpat300) and will be compared between both arms
Percentage of saturation <70% | First postoperative night
  will be measured by a home sleep study device (Watchpat300) and will be compared between both arms
Time (minutes) of saturation <90% | First postoperative night
  will be measured by a home sleep study device (Watchpat300) and will be compared between both arms
Time (minutes) of saturation <88% | First postoperative night
  will be measured by a home sleep study device (Watchpat300) and will be compared between both arms
Time (minutes) of saturation <85% | First postoperative night
  will be measured by a home sleep study device (Watchpat300) and will be compared between both arms
Time (minutes) of saturation <80% | First postoperative night
  will be measured by a home sleep study device (Watchpat300) and will be compared between both arms
Time (minutes) of saturation <70% | First postoperative night
  will be measured by a home sleep study device (Watchpat300) and will be compared between both arms
Total sleep time (minutes) | First postoperative night
  Total sleep time will be measured by a home sleep study device (Watchpat300) and will be compared between both arms
Percentage of REM sleep in total sleep time | First postoperative night
  Percentage of REM sleep will be measured by a home sleep study device (Watchpat300) and will be compared between both arms
Percentage of Deep sleep in total sleep time | First postoperative night
  Percentage of Deep sleep will be measured by a home sleep study device (Watchpat300) and will be compared between both arms
Percentage of light sleep in total sleep time | First postoperative night
  Percentage of light sleep will be measured by a home sleep study device (Watchpat300) and will be compared between both arms
Percentage of awake time | First postoperative night
  Percentage of awake time will be measured by a home sleep study device (Watchpat300) and will be compared between both arms

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hazebroek, Prof.dr., Principal Investigator — Rijnstate Hospital
Locations (1):
- Vitalys, Elst, Netherlands

IPD SHARING:
Plan to Share IPD: No